CLINICAL TRIAL: NCT04987801
Title: Evaluation of Drug Overdose Poisoning Cases and Indications for ICU Admission
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Peter Eissa Saad, Demonstrator at Forensic and clinical toxicology department, Assiut University
Other Study IDs: Drug overdose Evaluation
Record Dates: First submitted 2021-07-07; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Drug Toxicity
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Drug Toxicity — Patients who took over dose of Drugs

SUMMARY:
1. Evaluation of drug overdose cases presented to Assiut university hospitals' adults and pediatric emergency departments (EDs) in one year period.
2. Evaluation the role of intensive care unit (ICU) admission in these cases and possible scoring system for common groups of drug overdose.

DETAILED DESCRIPTION:
Poisoning is a medical emergency representing a health problem all over the world with an incidence rate that is variable from one place to another.

The nature of poison used varies in different parts of the world and may vary even in different parts of the same country.

The pattern of poisoning within a country depends on several factors such as the accessibility of various poisons, socio-economic status of the population, religious and cultural influences and drug prescription manners.

Drug overdose continues to be the most common cause of acute poisoning all over the world. An estimated 2 to 5 million poisonings and drug overdoses occur annually in the United States of America.

Overdose is the most common manifestation of deliberate self-harm behavior, and is a common cause of presentation to hospital Emergency Departments (EDs). It starts to get global attention due to its higher rate of morbidity and mortality in spite of being a preventable cause of death.

Acute drug overdosing is an important cause of organ dysfunction and metabolic derangements and the patients often require intensive care admission. Among patients admitted to hospital following drug overdoses, approximately 13-22% will require Intensive Care Unit (ICU) admission. Overdoses have been reported to account for 3.8-13.8% of all ICU admissions with 79.5-84% requiring mechanical ventilation in Australia.

The treatment and complications of patients with acute drug intoxication in ICU vary according the nature of the substance ingested, individual amount of drug, and the concomitant use of other substances. The interventions requiring critical care in acute drug-poisoned patients include the need for airways protection and mechanical ventilation, hemodynamic stabilization and needs for vasopressors, and specific procedures that would enhance the clearance of the toxins involved.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted or transferred to Assiut university hospitals' adults and pediatric EDs, with history of drug overdose intoxication within 24 hours prior to admission (single or multiple drug ingestions).
* Patients admitted or transferred to Assiut university hospitals' adults and pediatric EDs, with clinical signs and symptoms of drug overdose intoxication on examination.
* Patients admitted or transferred to Assiut university hospitals' adults and pediatric EDs, with blood and/or urine toxicology screens demonstrated the presence of non-prescribed, illicit drugs or inappropriately elevated levels of prescribed or over the-counter medications.

Exclusion Criteria:

* Patients admitted or transferred to Assiut university hospitals' adults and pediatric EDs, with history of drug overdose intoxication more than 24 hours.
* Patients admitted or transferred to Assiut university hospitals' adults and pediatric EDs, with history of non-drug intoxication, e.g insecticides poisoning

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who took over dose of Drugs
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of drug overdose cases presented to Assiut university hospitals' adults and pediatric E.D. | One year
  A) Sheet includes the following items:-
  1. Demographic data:
     Gender, Age, Marital status, Residence, Occupation, Special habits: smoking, drug abuse.
  2. Data regarding overdosed drug:
     Type, form, dose and method of administration and mode of exposure
  3. Symptoms of intoxication. B) Complete clinical examination
  C) Investigations:
  1. Routine: ABG, ECG, Electrolytes
  2. Specific Drug level, drug screening test in urine

SECONDARY OUTCOMES:
Evaluation of the indications of intensive care unit (ICU) admission in drug overdose cases. | one year
  Evaluation the role of intensive care unit (ICU) admission in drug overdose cases and possible scoring system for common groups of drug overdose:
  Patients admitted to ICU will be monitored regarding:
  * Criteria of admission: acid base disturbance, altered conscious level, organ failure, etc.
  * Intervention methods: mechanical ventilation, inotropes, dialysis, etc.
  * Period of ICU Admission.
  * Fate : complete recovery, complications, death

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Asyut, Egypt

REFERENCES:
- [Background] Athavale V, Green C, Lim KZ, Wong C, Tiruvoipati R. Characteristics and outcomes of patients with drug overdose requiring admission to Intensive Care Unit. Australas Psychiatry. 2017 Oct;25(5):489-493. doi: 10.1177/1039856217706824. Epub 2017 Jul 13. PMID 28703691
- [Background] Bakhaidar M, Jan S, Farahat F, Attar A, Alsaywid B, Abuznadah W. Pattern of drug overdose and chemical poisoning among patients attending an emergency department, western Saudi Arabia. J Community Health. 2015 Feb;40(1):57-61. doi: 10.1007/s10900-014-9895-x. PMID 24927975
- [Background] Jayakrishnan B, Al Asmi A, Al Qassabi A, Nandhagopal R, Mohammed I. Acute drug overdose: clinical profile, etiologic spectrum and determinants of duration of intensive medical treatment. Oman Med J. 2012 Nov;27(6):501-4. doi: 10.5001/omj.2012.120. PMID 23226824
- [Background] Savage M, Kung R, Green C, Thia B, Perera D, Tiruvoipati R. Predictors of ICU admission and long-term outcomes in overdose presentations to Emergency Department. Australas Psychiatry. 2020 Feb;28(1):75-79. doi: 10.1177/1039856219889317. Epub 2020 Jan 8. PMID 31912753
- [Background] Tawfik, H., & Khalifa, E. (2017). Evaluation of Poisoning and Drug Overdose among Cases Presented to Poison Control Centre, Ain Shams University Hospital during the Year 2015. Ain Shams Journal of Forensic Medicine and Clinical Toxicology, 29(2), 100-112.
- [Background] Zhao M, Ji XP, Wang NN, Liu SY, Wang YZ. Study of poisoning pattern at China Medical University from 1997 to 2007. Public Health. 2009 Jun;123(6):454-5. doi: 10.1016/j.puhe.2009.04.010. Epub 2009 Jun 3. No abstract available. PMID 19497600
- [Background] Cioccari L, Luethi N, Bailey M, Pilcher D, Bellomo R. Characteristics and outcomes of critically ill patients with drug overdose in Australia and New Zealand. Crit Care Resusc. 2017 Mar;19(1):14-22. PMID 28215127
- [Background] Orsini, Jose, et al.